CLINICAL TRIAL: NCT01355965
Title: Phase 1 Clinical Trial of Autologous Mesothelin Re-Directed T Cells Administered Intravenously in Patients With Progressive Malignant Pleural Mesothelioma
Brief Title: Autologous Redirected RNA Meso-CIR T Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 17510
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: completed standard first line therapy; platinum based double regimen; Progressive Disease; chosen not to pursue primary standard of care therapy
MeSH Terms: conditions — Mesothelioma, Malignant; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 - One dose of cells (Experimental): Subjects receive one dose of 1x108 cells on day 0 followed by one dose of 1x109 autologous transfected anti-mesothelin CAR T cells on day 7.
  Interventions: Biological: Autologous T cells
- Cohort 2 - three doses of cells (Experimental): receive three doses of 1x108 cells on day 0, 2, 4 (Monday-Wednesday-Friday (MWF) of Cycle 1) followed by three doses of 1x109 T cells on day 7, 9, 11 (MWF of Cycle 2). Total target dose for Cohort 2 is 3.3x109 cells.
  Interventions: Biological: Autologous T cells

INTERVENTIONS:
Biological: Autologous T cells

SUMMARY:
To determine the safety and manufacturing feasibility of IV autologous chimeric immune receptor (CIR) T cells transfected with anti-mesothelin messenger RNA (mRNA) expressing a single chain antibody variable fragment linked to the intracellular CD 3 zeta T cell receptor domain and the 4-1BB costimulatory domain.

DETAILED DESCRIPTION:
The purpose of this study is to test the safety of infusing the study product CIR T cells. These T cells are made using T cells obtained through apheresis and introducing the T cells to a temporary gene which will cause them to start making a new type of antibody that will attach mesothelin (this antibody is found on the surface of the cancer cells). In theory, once the modified T cells attach to mesothelin, the cells will be activated to stimulate the subject's own immune system to attack the mesothelin cells. This type of modified cell is called a T cell transduced transfected with chimeric anti-mesothelin immunoreceptor. Subjects will be enrolled serially with all subjects receiving 1xe8 to 1x1e9 modified CIR T cells every other day for 3 infusions. Each patient will be observed for 9 days for toxicity assessment prior to receiving a second cycle of modified CIR T cells every other day for 3 infusions. The preceding subject must have completed the two-cycle regimen and been observed for toxicity through day 21 before the next subject can be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed MPM (epithelial or biphasic).
* Subjects must have completed standard first line therapy with a platinum-based double regimen and had PD or they must have chosen not to pursue primary standard of care therapy.
* ECOG performance status 0 to 1.
* Age greater than 18 years
* Life expectancy > 4 months
* At least 2 weeks since prior and no other concurrent chemotherapy, radiotherapy, or immunotherapy (e.g., interferons, tumor necrosis factor, interleukins, or monoclonal antibodies). In addition, the patient must have fully recovered from any adverse events related to these agents.
* More than 4 weeks since prior and no other concurrent investigational agents.
* Subjects must have measurable disease as defined by accepted MPM measurement techniques (modified RECIST criteria).
* Blood coagulation parameters: PT such that international normalized ratio (INR) is < 1.5 (or an in-range INR, usually between 2 and 3, if a subject is on a stable dose of therapeutic warfarin for management of venous thrombosis including pulmonary thromboembolus) and a PTT < 1.2 times the upper limit of normal.
* Subjects must have adequate venous peripheral access for apheresis. Patients must also have adequate venous access for subsequent modified CIR T-cell administration which can be done through a central venous access (e.g. port of systemic chemotherapy).
* Short-term therapy for acute conditions not specifically related to MPM is allowed if such therapy does not include any immune modulating agents.
* Male and Female subjects agree to use approved contraceptive methods (e.g. birth control pills, barrier device, intrauterine device , abstinence) during the study and for 3 months following the last dose of the study cell infusion.
* Subject must understand and sign the study-specific informed consent .
* Satisfactory organ and bone marrow function as defined by :

Absolute neutrophil count > 1,000/µl Platelets > 100,000/µl Hematocrit > 30 % AST(SGOT)/ALT(SGPT) < 3x the institutional normal upper limit Bilirubin < 2.0 mg/dL unless secondary to malignant bile duct obstruction Creatinine < 1.5x the institutional normal upper limit

Exclusion Criteria:

* Previously treated with any investigation therapy within 1 month prior to screening.
* Sacromatoid MPM histology which does not express mesothelin
* Prior invasive malignancies unless surgically and medically cured without evidence of recurrent disease for 5 years with the exception of non-melanoma skin cancer, prostate cancer with PSA level < 1.0.
* Prior hematologic malignancy with bone marrow transplantation or immune modifying therapy within the past 4 weeks with the exception of thyroid replacement.
* Use of immunosuppressive drugs with 4 weeks prior to study entry, or anticipated use of immunosuppressive agents.
* Any clinically -significant pericardial effusion, CHF (NY Heart Association Grade II-IV ), or cardiovascular condition.
* Any clinically -significant pleural effusion or ascites that cannot be drained with standard approaches or with pre-enrollment in dwelling drainage device placement.
* Forced vital capacity < 50% predicted, DLCO < 40% predicted.
* Underlying lung disease requiring supplemental oxygen therapy.
* Have a recognized immunodeficiency disease including cellular immunodeficiency, hypogammaglobulinemia, or dysgammaglobulinemia; patients who have acquired hereditary, congenital immunodeficiency.
* Viral infections: HIV, HCV, HBV.
* Pregnant women are excluded from this study because autologous transduced T cells, breastfeeding should be discontinued if the mother is treated.
* Feasibility assessment during screening demonstrates < 30% transfection of target lymphocytes, or < 5-fold expansion in modified CIR T-cells in response to CD3/CD28 costimulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-05; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Until week 4
  Occurence of study related adverse events greater than to equal to Grade 3 events that are possibly, likely or definitely related to study treatment.

SECONDARY OUTCOMES:
Clinical response Rate | through 6 months post dosing
  Effect of CIR T cell infusion on systemic adaptive and innate immunity

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Haas, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Maus MV, Haas AR, Beatty GL, Albelda SM, Levine BL, Liu X, Zhao Y, Kalos M, June CH. T cells expressing chimeric antigen receptors can cause anaphylaxis in humans. Cancer Immunol Res. 2013 Jul;1(1):26-31. doi: 10.1158/2326-6066.CIR-13-0006. Epub 2013 Apr 7. PMID 24777247